CLINICAL TRIAL: NCT06309953
Title: An Open-Label, Multicenter, Phase 4 Study to Evaluate Early Treatment Outcomes With Miebo™ in Subjects With Dry Eye Disease
Brief Title: A Study to Evaluate Early Treatment Outcomes With Miebo™ in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 937
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — perfluorohexyl-octan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Miebo treatment (Experimental)
  Interventions: Drug: Miebo

INTERVENTIONS:
Drug: Miebo — Miebo® (perfluorohexyloctane ophthalmic solution) Dosage: one drop of MIEBO four times daily into each eye Dosage form: Ophthalmic solution: 100% perfluorohexyloctane. Frequency: 4 times daily for 14 days

SUMMARY:
An Open-Label, Multicenter, Phase 4 Study to Evaluate Early Treatment Outcomes With Miebo™ in Subjects With Dry Eye Disease

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate early outcomes with Miebo treatment in subjects with Dry Eye Disease (DED)

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of consent
2. Able to provide written voluntary informed consent
3. The same eye must satisfy the below inclusion criteria (a-e):

   1. Subject-reported history of DED in at least 1 eye for at least 6 months prior to Visit 1
   2. Tear-film break-up time ≤5 seconds at Visit 1
   3. Total corneal fluorescein staining score ≥4 and ≤11 (ie, sum of inferior, superior, central, nasal, and temporal) according to the National Eye Institute scale at Visit 1
   4. Total meibomian gland dysfunction score ≥3 (range, 0-15)
   5. Unanesthetized Schirmer's test I score ≥5 mm
4. Ocular Surface Disease Index (OSDI) ≥25 at Visit 1
5. Able and willing to follow instructions, including participation in all trial assessments and visits.

Exclusion Criteria:

Note: Ocular exclusion criteria are relevant to both eyes, such that meeting a criterion in either eye excludes the subject from the study

1. Had received Miebo as a prescription or as a study treatment in previous Miebo clinical studies
2. Have any clinically significant ocular surface slit lamp findings at Visit 1 and/or, in the opinion of the Investigator, have any findings that could interfere with trial parameters, including:

   1. History of eye trauma
   2. History of Stevens-Johnson syndrome
   3. Active blepharitis or lid margin inflammation
   4. DED secondary to scarring, irradiation, alkali burns, cicatricial pemphigoid, or destruction of conjunctival goblet cells (as with vitamin A deficiency)
   5. Abnormal lid anatomy causing incomplete eyelid closure
   6. Abnormal cornea shape (keratoconus)
   7. Corneal epithelial defect or significant confluent or filaments
   8. History of herpetic keratitis
   9. Pterygium
   10. Ocular or periocular rosacea
3. Use of any of the following ocular therapies within 60 days prior to Visit 1: Vuity®, any topical ocular steroid treatments, prescription dry eye therapy including varenicline nasal spray, or topical anti-glaucoma medication
4. Had a LipiFlow® procedure, intense pulse light procedure, or any kind of other procedure affecting meibomian glands within 6 months prior to Visit 1
5. Had received or removed a permanent punctum plug within 3 months (6 months for dissolvable plugs) prior to Visit 1
6. Use of any eye drops (prescription or over-the counter, such as artificial tears or Lumify®) and/or TrueTear™ device (intranasal tear neurostimulator) within 24 hours prior to Visit 1
7. Have active ocular allergies or ocular allergies that are expected to be active during the trial period.
8. Have worn contact lenses within 1 month prior to Visit 1 or planned wear during the study.
9. Have undergone intraocular surgery or ocular laser surgery within 3 months prior to Visit 1; have undergone refractive surgery within 2 years prior to Visit 1
10. Have active ocular or systemic infection (bacterial, viral, or fungal), including fever.
11. Female subjects who are pregnant, nursing, or planning a pregnancy
12. Female subjects of childbearing potential who are not using an acceptable means of birth control; acceptable methods of contraception include hormonal (oral, implantable, injectable, or transdermal) contraception; mechanical (spermicide in conjunction with a barrier such as a diaphragm or condom) contraception; intrauterine device; or surgical sterilization of partner. For non-sexually active female subjects, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the trial, she must agree to use adequate birth control as defined above for the remainder of the trial.
13. Have an uncontrolled systemic disease that, in the opinion of the Investigator, will interfere with the trial
14. Have a known allergy and/or sensitivity to the study treatment
15. Use of any oral medications known to cause ocular drying (eg, antihistamines, antidepressants, etc.) on a non-stable regimen within 1 month prior to Visit 1 or is expected to be unstable during the trial
16. Have taken isotretinoin (eg, Accutane, Myorisan, Claravis, Amnesteem) within 6 months prior to Visit 1
17. Have corrected visual acuity (VA) worse than or equal to +0.7 logarithm of the minimum angle of resolution (logMAR), as assessed with Snellen chart at Visit 1
18. Are currently enrolled in an investigational drug or device study or had used an investigational drug or device within 60 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Site 207, Birmingham, Alabama
  - Site 205, Petaluma, California
  - Site 203, Pittsburg, Kansas
  - Site 204, Stillwater, Minnesota
  - Site 202, Kansas City, Missouri
  - Site 201, Brecksville, Ohio
  - Site 206, Westlake, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bacharach J, Kannarr SR, Verachtert A, Gupta PK, Razeen M, Cavet ME, Vittitow JL, Lang J, Chester TM, Ziemanski JF, White DE. Early Effects of Perfluorohexyloctane Ophthalmic Solution on Patient-Reported Outcomes in Dry Eye Disease: A Prospective, Open-Label, Multicenter Study. Ophthalmol Ther. 2025 Apr;14(4):693-704. doi: 10.1007/s40123-025-01097-z. Epub 2025 Feb 22. PMID 39985746

RESULTS

PARTICIPANT FLOW:
Groups:
- Miebo Treatment: Intervention: Miebo® (perfluorohexyloctane ophthalmic solution) Dosage: one drop of MIEBO four times daily into each eye Dosage form: Ophthalmic solution: 100% perfluorohexyloctane. Frequency: 4 times daily for 14 days
Period: Overall Study
Arm/Group | Miebo Treatment
Started | 99
Completed | 98
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Miebo Treatment: Miebo: Miebo treatment
Arm/Group | Miebo Treatment
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 90
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 99

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (CFB) in Dry Eye Symptom Severity at Visit 3
Description: Mean change from baseline (CFB) in dry eye symptom severity at Visit 3 (Day 7 ± 1 day) Scale name: Visual Analog Scale Range: min: 0%, max: 100%; 0% corresponds to "none" and 100% corresponds to "worst severity possible" Intrepretation: VAS is a subjective measurement tool that consists of a horizontal assessment line, of 100 mm (10 cm) length where patients place a vertical mark to indicate the level of perceived severity of symptoms. Higher values indicate worse disease severity, lower values indicate better outcome with treatment
Time Frame: Change from baseline in VAS at Visit 3 (Day 7 ± 1 day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Miebo Treatment
Number analyzed (Participants) | 99
score on a scale | -44.5 (25.15)

ADVERSE EVENTS:
Time Frame: Assessed for approximately 3.5 months
Arm/Group | Miebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT06309953/Prot_SAP_000.pdf